CLINICAL TRIAL: NCT01930266
Title: Young Adults With Life Threatening Cow's Milk Allergy: Risks of Decrease Bone Mineralization and Methods of Calcium Supplementation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Helsinki commitee, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 187/11
Record Dates: First submitted 2013-08-25; First posted 2013-08-28 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Bone Mineral Density in Cow's Milk Allergic Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Observational (No Intervention): Patients will receive general dietary instructions with an annual follow-up. At this follow up, a repeat BMD, dietary and laboratory evaluation will be performed.
- Interventional. (Active Comparator): Patients will receive detailed dietary instructions with periodic (3 month) follow up. At the follow-up patients will be assessed whether they reached their calcium intake goals both quantitatively and whether appropriate calcium sources were utilized.
  Interventions: Behavioral: Active comparator
- Active interventional (Experimental): Patients will receive detailed dietary instructions and active follow up with diary and email reports. Inclusion in group C will be predicated upon intake of 100% DRI of calcium primarily by food sources, with the addition of Calcium Carbonate 600 mg, if necessary
  Interventions: Dietary Supplement: Experimental

INTERVENTIONS:
Dietary Supplement: Experimental
  Arms: Active interventional
Behavioral: Active comparator
  Arms: Interventional.

SUMMARY:
Diet is the only source for calcium and the most important dietary source are dairy products. This presents a difficulty for children with IgE-mediated cow's milk allergy, who are unable to consume milk. We noted that IgE-CMA allergic young adults have a significant decrease in bone mineral density (BMD) compared to international reference values and also to geographically and age matched normal controls.

Working hypothesis: Young adults with IgE-CMA have significantly lower BMD than age and gender matched controls. This can be reversed by introducing dairy products following recovery from allergy, or by enriching the diet via other calcium sources.

DETAILED DESCRIPTION:
The aims of the study are 1. To study the prevalence and severity of reduced BMD among IgE-CMA allergy patients 2. to estimate the potential of recovery from reduced BMD after administration of milk during oral immunotherapy.

3. To determine the efficacy of intervention with other (non-dairy) calcium enriched diets in IgE-CMA young adults, utilizing several methods to direct compliance.

Methods: We will study the bone mineral content (BMC), BMD, serum values of bone turnover factor, dietary and lifestyle questionnaires of 150 post pubertal IgE-CMA patients with no history of dairy consumption and 150 age and gender matched normal controls. Separately, we will compare the above values of these patients to those of former IgE-CMA patients who now ingest milk after recovery from allergy. Finally, we will examine the effects of including non-dairy dietary sources of calcium in IgE-CMA patients, with different groups receiving different degrees of interventional guidance.

The study will provide insight into the bone health of CMA patients, and provide guidance as to effective dietary treatments and its implementation. Furthermore, important nutritional data on the best methods for intervention to reduce osteoporosis will likely be learnt, that should have far reaching ramifications, not only to this particular population, but to osteoporosis patients, at large.

ELIGIBILITY:
Inclusion Criteria:

All post pubertal males and females diagnosed with IgE-mediated CMP allergy were eligible Puberty in both sexes was determined by signs of Tanner stage IV. Females were at least two years after menarche The minimal age for girls was 16 years and for boys 17.5 years old. The maximal age to be included in this study was 30 years old

Exclusion Criteria:

female's history of pregnancy, and in both genders any 128 bone affecting disease/treatment, systemic steroid treatment for a period longer than 4 weeks or multiple short courses of systemic steroid treatments.

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
efficacy of calcium supplemetation in preventing BMD loss in cow's milk allergic patients | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Asaf Harofeh Medical Center, Beer Yaakov, Zerifin, Israel